CLINICAL TRIAL: NCT03642847
Title: A PHASE 1B, RANDOMIZED, CONTROLLED, DOUBLE-BLIND TRIAL TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF MULTIVALENT PNEUMOCOCCAL CONJUGATE VACCINES IN HEALTHY JAPANESE ADULTS 18 TO 49 YEARS OF AGE
Brief Title: Trial to Evaluate the Safety and Immunogenicity of Multivalent Pneumococcal Vaccines in Japanese Adults 18 to 49 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B7471005
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Prevnar 13 (Active Comparator): 13 valent Pneumococcal Conjugate
  Interventions: Biological: Prevnar 13
- multivalent pneumococcal conjugate formulation 1 (Experimental): multivalent pneumococcal conjugate formulation 1
  Interventions: Biological: multivalent pneumococcal conjugate formulation 1
- multivalent pneumococcal conjugate formulation 2 (Experimental): multivalent pneumococcal conjugate formulation 2
  Interventions: Biological: multivalent pneumococcal conjugate formulation 2

INTERVENTIONS:
Biological: Prevnar 13 — 13 valent Pneumococcal Conjugate
  Arms: Prevnar 13
Biological: multivalent pneumococcal conjugate formulation 1 — multivalent pneumococcal conjugate formulation 1
  Arms: multivalent pneumococcal conjugate formulation 1
Biological: multivalent pneumococcal conjugate formulation 2 — multivalent pneumococcal conjugate formulation 2
  Arms: multivalent pneumococcal conjugate formulation 2

SUMMARY:
This Phase 1b will describe the safety and immunogenicity of 2 multivalent pneumococcal conjugate vaccine formulations in healthy Japanese adults in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Japanese subjects 18 to 49 years of age, defined as Japanese born in Japan, with both parents and 4 grandparents who wer born in Japan (family tree by history), and who have not lived outside of Japan for more than 5 years total (confirmed by passport or interview)

Exclusion Criteria:

* Participation in other studies involving investigational drug(s), investigational vaccines, or investigational medical devised within 28 days prior to study entry and/or during study participation. Participation in purely observational studies is acceptable.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Subjects reporting prompted local reactions within 14 days after vaccination (redness, swelling, and pain at the injection site). | 14 days after vaccination
  Subjects reporting prompted local reactions within 14 days after vaccination (redness, swelling, and pain at the injection site).
Subjects reporting prompted systemic events within 14 days after vaccination (fever, headache, fatigue, muscle pain, and joint pain). | 14 days after vaccination
  Subjects reporting prompted systemic events within 14 days after vaccination (fever, headache, fatigue, muscle pain, and joint pain).
Subjects reporting adverse events (AEs) within 1 month after vaccination. | 1 month after vaccination
  Subjects reporting adverse events (AEs) within 1 month after vaccination.
Subjects reporting serious adverse events (SAEs) within 6 months after vaccination. | 6 months after vaccination
  Subjects reporting serious adverse events (SAEs) within 6 months after vaccination.
Subjects reporting newly diagnosed chronic medical conditions (NDCMCs) within 6 months after vaccination. | 6 months after vaccination
  Subjects reporting newly diagnosed chronic medical conditions (NDCMCs) within 6 months after vaccination.

SECONDARY OUTCOMES:
Immunogenicity | 1 month after vaccination
  Pneumococcal serotype-specific OPA titers 1 month after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Collaborative Neuroscience Network, LLC., Garden Grove, California
  - Collaborative Neuroscience Network, LLC., Long Beach, California
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Clinilabs Drug Development Corporation, Eatontown, New Jersey

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Fitz-Patrick D, Young M Jr, Scott DA, Scully IL, Baugher G, Peng Y, Jansen KU, Gruber W, Watson W. A randomized phase 1 study of the safety and immunogenicity of 2 novel pneumococcal conjugate vaccines in healthy Japanese adults in the United States. Hum Vaccin Immunother. 2021 Jul 3;17(7):2249-2256. doi: 10.1080/21645515.2020.1863177. Epub 2021 Feb 5. PMID 33545022
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7471005&StudyName=A+PHASE+1B%2C+RANDOMIZED%2C+CONTROLLED%2C+DOUBLE-BLIND+TRIAL+TO+EVALUATE+THE+SAFETY+AND+IMMUNOGENICITY+OF+MULTIVALENT+PNEUMOCOCCAL+CONJUGATE+VACCINES+IN+HEALTHY+JAPANESE+ADULTS+18+TO+49+YEARS+OF+AGE